CLINICAL TRIAL: NCT03169231
Title: A Phase 2b, Randomized, Blinded and Placebo-Controlled Trial to Evaluate the Safety and Efficacy of Longeveron Allogenic Human Mesenchymal Stem Cells Infusion in Patients With Aging Frailty
Brief Title: Phase IIb Trial to Evaluate Longeveron Mesenchymal Stem Cells to Treat Aging Frailty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Longeveron Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 001-03
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Aging Frailty

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Study Group A (Experimental): Single peripheral IV infusion of 25 million Longeveron Mesenchymal Stem Cells (LMSCs)
  Interventions: Biological: Longeveron Mesenchymal Stem Cells (LMSCs)
- Study Group B (Experimental): Single peripheral IV infusion of 50 million Longeveron Mesenchymal Stem Cells (LMSCs)
  Interventions: Biological: Longeveron Mesenchymal Stem Cells (LMSCs)
- Study Group C (Experimental): Single peripheral IV infusion of 100 million Longeveron Mesenchymal Stem Cells (LMSCs)
  Interventions: Biological: Longeveron Mesenchymal Stem Cells (LMSCs)
- Study Group D (Experimental): Single peripheral IV infusion of 200 million Longeveron Mesenchymal Stem Cells (LMSCs)
  Interventions: Biological: Longeveron Mesenchymal Stem Cells (LMSCs)
- Study Group E (Placebo Comparator): Single peripheral IV infusion of placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Longeveron Mesenchymal Stem Cells (LMSCs) — Intravenously delivered
  Arms: Study Group A; Study Group B; Study Group C; Study Group D
Other: Placebo — Intravenously delivered
  Arms: Study Group E

SUMMARY:
This is a randomized, placebo-controlled, double-blind, parallel arm, multi-center Phase 2b study.

DETAILED DESCRIPTION:
The objectives of this study are to assess safety and efficacy of Longeveron Mesenchymal Stem Cells (LMSCs) compared to placebo on 1) functional mobility and exercise tolerance, 2) patient-reported physical function, and 3) the inflammatory cytokine biomarker tumor necrosis factor (TNF-alpha).

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent and comply with all procedures required by the Protocol.
2. Be >70 and < 85 years of age at the time of signing the Informed Consent Form.
3. Have a Canadian Study on Health and Aging (CSHA) Clinical Frailty Scale score of 5 "mildly frail" or 6 "moderately frail".
4. Have a 6 minute walk distance of > 200m and < 400 m. Distances of two 6MWTs are to be within 15% of each other.
5. Have a serum TNF-alpha level > 2.5 pg/mL

Exclusion Criteria:

1. Be unwilling or unable to perform any of the assessments required by the protocol.
2. Have a diagnosis of any disabling neurologic disorder, including, but not limited to, Parkinson's disease, Amyotrophic Lateral Sclerosis, multiple sclerosis, cerebrovascular accident with residual deficits (e.g., muscle weakness or gait disorder), or diagnosis of dementia.
3. Have a score of 24 or lower on the Mini Mental State Examination (MMSE)
4. Have poorly controlled blood glucose levels (HbA1c >8.0%).
5. Have a clinical history of malignancy within 2.5 years (i.e., subjects with prior malignancy must be cancer free for 2.5 years) except curatively-treated basal cell carcinoma, melanoma in situ or cervical carcinoma.
6. Have any condition that in the opinion of the Principal Investigator limits lifespan to < 1 year.
7. Have autoimmune disease (e.g. rheumatoid arthritis, systemic lupus erythematosus).
8. Be using chronic immunosuppressant therapy such as high-dose corticosteroids or TNF-alpha antagonists (prednisone use at doses of < 5 mg daily is allowed).
9. Test positive for hepatitis B virus

   a. If the subject tests positive for anti-hepatitis B core antigen (HBc) or anti-HBs, they must be currently receiving treatment for Hepatitis B prior to infusion and remain on treatment throughout the study.
10. Test positive for verimic Hepatitis C virus, HIV1/2, or syphilis
11. Have a resting blood oxygen saturation of <93% (measured by pulse oximetry).
12. Known or suspected alcohol or drug abuse within three years preceding Screening
13. Have a known hypersensitivity to dimethyl sulfoxide (DMSO).
14. Be an organ transplant recipient (other than transplantation for corneal, bone, skin, ligament, or tendon).
15. Be actively listed (or expected future listing) for transplant of any organ (other than corneal transplant).
16. Have any clinically important abnormal screening laboratory values, including, but not limited to:

    1. Hemoglobin <10.0 g/dL,
    2. White blood cell <2,500/ul, or platelet count <100,000/ul
    3. Liver dysfunction evidenced by enzymes (AST and ALT) > 3 times the upper limit of normal (ULN)
    4. Coagulopathy (INR>1.3) not due to a reversible cause (e.g. warfarin and/or Factor Xa inhibitors).
17. Uncontrolled hypertension (resting systolic blood pressure >180 mm Hg or diastolic blood pressure of > 110 mm Hg at Screening)
18. Have unstable angina pectoris, uncontrolled or severe peripheral artery disease within the previous 3 months.
19. Have congestive heart failure defined by NYHS (New York Heart Association) Class III or IV, or an ejection fraction of <25%.
20. Have a coronary artery bypass surgery, angioplasty, or peripheral vascular disease revasculation or a myocardial infarction within previous 3 months.
21. Have severe pulmonary dysfunction: acute exacerbation of chronic obstructive lung disease stage III or IV (Gold classification), and/or PaO2 levels <60 mmHg.
22. Have a partial ileal gastric bypass, or other significant intestinal malabsorption.
23. Have advanced liver or renal disease
24. Have cognitive or language barriers that prohibit obtaining informed consent or any study elements.
25. Be currently hospitalized, or living in an assisted living facility or a long-term care facility.
26. Be currently participating (or participated within the previous 30 days of consent) in an investigational therapeutic or device trial.
27. Have a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study, or interfere with the patient's participation for the full duration of the study.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 6 Minute Walk Test (6MWT) compared to placebo | Baseline and 180 days post-infusion
  Change from baseline in 6MWT compared to placebo at 180 days post-infusion

SECONDARY OUTCOMES:
Change in patient reported outcome of overall physical function capacity using the PROMIS-Physical Function-Short Form 20a compared to placebo | 180 days post-infusion
  Change from baseline in physical function will be measured to assess Patient-Reported Outcome Measurement compared to placebo at 180 days post infusion.
Change in TNF-alpha compared to placebo | 180 days post-infusion
  Change in serum TNF-alpha compared to placebo

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Soffer Health Institute, Aventura, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Miami VA Healthcare System, Miami, Florida
  - Vista Health Research, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Advanced Research for Health Improvement, LLC, Naples, Florida

IPD SHARING:
Plan to Share IPD: No